CLINICAL TRIAL: NCT00464451
Title: Prospective, Double Blinded,Randomized Controlled Trial of Dexmedetomidine Versus Chloral Hydrate for Pediatric Sedation During EEG
Brief Title: Dexmedetomidine Versus Chloral Hydrate for Pediatric Sedation During EEG
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain approval from FDA for use of chloral hydrate
Sponsor: Wesley Medical Center (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Lindall E.Smith, Medical Doctor, Wesley Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dex for Ped EEG
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Procedural Sedation
MeSH Terms: interventions — Dexmedetomidine; Chloral Hydrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dexmedetomidine sedated pediatric patients undergoing EEG study.
  Interventions: Drug: Dexmedetomidine
- 2 (Active Comparator): Chloral hydrate sedated pediatric patients undergoing sedated EEG study.
  Interventions: Drug: Chloral hydrate

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 3 micrograms per kilogram per os; subsequent dose of 1 microgram per kilogram per os if necessary to treat inadequate sedation 30 minutes following initial dosing.
  Arms: 1
Drug: Chloral hydrate — Chloral hydrate 75 milligrams per kilogram per os; subsequent dose of 25 milligrams per kilogram per os if necessary to treat inadequate sedation 30 minutes following initial dosing.
  Arms: 2

SUMMARY:
The purpose of the study is:

1. To compare the efficacy of dexmedetomidine versus chloral hydrate as pediatric sedation agents for EEG studies. Efficacy will be determined by successful EEG study completion and by minimum degree of sedation induced patient agitation (SAS score).
2. To compare the safety and adverse event profile of dexmedetomidine versus chloral hydrate during sedation of pediatric patients for EEG studies. Comparison will be based on variance of vital signs (HR, MAP, RR, O2SAT, ETCO2) from baseline during sedation as well as the frequency of adverse events during and following sedation.
3. To compare quality of EEG recording obtained with dexmedetomidine or chloral hydrate and to those of non-sedated pediatric EEG studies. Quality will be determined by the degree of background beta-wave activity.

DETAILED DESCRIPTION:
Pediatric patients undergoing EEG studies often require sedation because of failure to stay still during recording of EEG (the difficulty in them obtaining a sleep state on their own during a specific time for the procedure). The ideal sedation agent (for an EEG) should have a rapid onset of action, moderate duration of effect, minimal or absent side-effect profile and a minimal or no effect on EEG quality. Historically, chloral hydrate has been the oral agent of choice for sedating pediatric patients for EEGs. However, chloral hydrate use has been fraught with many problems such as sedation failure, drug-enhanced background beta-wave activity affecting EEG quality, and (especially in pediatric patients) an unpleasant intoxicated-like experience while recovering from sedation. Uncommon but specific adverse events associated with the use of chloral hydrate include gastric irritation causing nausea, vomiting, diarrhea; residual sleepiness or "hangover"; rashes, fever, dizziness, ataxia; disorientation, paradoxical excitement, and respiratory depression (especially when combined with other sedatives or narcotics). Side effect profile and drug interference in EEG quality of chloral hydrate necessitates looking for alternate agent for EEG sedation. Clonidine has been shown to have better safety profile and lack of drug effect on EEG quality in Autistic children when compared to chloral hydrate. The beneficial effects of clonidine have been ascribed to its alpha-2 receptor agonist activity. We believe new alpha-2 agonist dexmedetomidine should have better safety profile with minimal or no effect in EEG quality because of its selective action on alpha-2 receptor.

Compared with clonidine, dexmedetomidine is more specific for the alpha-2 receptor and has a shorter elimination half-life. It produces dose-dependent sedation, anxiolysis and analgesia without respiratory depression.

Dexmedetomidine produces an unusually cooperative form of sedation, in which patients easily transition from sleep to wakefulness and then back to sleep when not stimulated. Its use is associated with less disinhibition than what has commonly been associated with other sedation agents like propofol and the benzodiazepines. Hemodynamic effects of dexmedetomidine result from peripheral and central mechanisms (peripheral vascular smooth muscle constriction, diminished central sympathetic outflow, and an increase in vagal activity) with a net result of significant reduction in circulating catecholamines, modest reduction in blood pressure, and a modest reduction in heart rate. Alpha-2 agonists have been shown to have minimal effects on ventilation in both healthy volunteers as well as in ICU patients. The benign effect of this class of drug on ventilatory drive is underscored by the approval of dexmedetomidine by the FDA as the only critical care sedative recommended for continuous use after extubation. Although alpha-2 agonists attenuate responses to stress, including neurohumoral responses, short term use of dexmedetomidine (<24 hours) does not significantly reduce serum cortisol levels. Bioavailability studies have demonstrated dexmedetomidine to be well absorbed systemically through the oral mucosa (up to 82 % compared to IV administration) and therefore, buccal dosing may provide an effective, noninvasive route to administer the drug. Orally administered dexmedetomidine has been successfully utilized as a pre-medication for pediatric procedural sedation or anesthetic induction to lessen anxiety and psychological impact of procedures with a dose range of 1-4.2 micrograms/kg (mean dose: 2.6 +/- 0.83 micrograms/kg). A large portion of the subjects in this study had neurobehavioral disorders and all were spontaneously breathing, non-intubated patients. None of the subjects experienced clinically significant changes in their cardiorespiratory parameters. Another study demonstrated successful sedation and analgesia is spontaneously breathing, non-intubated post-cardiothoracic surgery patients (ages 1 month to 21 years of age) with IV infusion of dexmedetomidine. No significant change in respiratory rate was noted. While several pediatric studies have explored the use of dexmedetomidine for post-operative and procedural sedation / analgesia in children with favorable results, it is not currently approved by the FDA for procedural sedation in children. Uncommon but specific adverse events associated with the use of dexmedetomidine include hypertension, hypotension, bradycardia, tachycardia, nausea, vomiting, fever, anemia, and hypoxia.

In summary, dexmedetomidine has the potential to be a good sedative agent for procedural and non procedural sedation in children, in part because of its favorable side-effect profile, minimal effect on respiratory drive, and minimal emergence agitation after the procedure. In addition, its sublingual bioavailability makes it attractive as an alternate oral agent for EEG sedation. It causes natural sleep; and because children may be intentionally aroused during its sedation and then resume sleep when not stimulated, it allows for complete EEG recordings containing awake, drowsy and sleep states.

We hypothesize that the use of dexmedetomidine for sedation in pediatric EEG studies will be more efficacious than chloral hydrate with a superior safety profile, patient tolerance and acceptance. We also hypothesize that the use of dexmedetomidine will minimize the degree of drug-enhanced background Beta-activity in sedated EEG recordings.

ELIGIBILITY:
Inclusion Criteria:

1. EEG study patients
2. Age less than 18 years
3. No contraindication for the use of chloral hydrate or dexmedetomidine

Exclusion Criteria:

1. Active, uncontrolled Gastroesophageal Reflux Disease (GERD)
2. Active, uncontrolled vomiting
3. Current history of apnea requiring apnea monitoring
4. Active, current respiratory issues that are different from the baseline status
5. Unstable cardiac status
6. Craniofacial anomaly with risk of inadequate bag-valve-mask ventilation
7. Current use of digoxin, betablockers, or calcium channel blockers
8. Current, active cerebral vascular disease
9. Patient treated with clonidine within the preceding one month
10. Prior history of drug reaction or sedation failure with either drug

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Sedation success with EEG study completion | 2 hours
Degree of sedation medication induces patient agitation. | 4 hours
Variance of vital signs from baseline during medication induced sedation for EEG study | 4 hours
Time to recovery from sedation. | 4 hours
Occurrence of adverse events. | 24 hours

SECONDARY OUTCOMES:
EEG record quality (degree of background beta-wave activity, levels of consciousness achieved, and degree of movement artifact) between sedated and non-sedated groups. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lindall E Smith, MD, Principal Investigator — University of Kansas School of Medicine-Wichita
Locations (1):
- Pediatric Sedation Unit, Wesley Medical Center, Wichita, Kansas, United States